CLINICAL TRIAL: NCT06935786
Title: SEDentary Lifestyle, Mortality and Major Adverse Clinical Outcomes in Chronic KIDney Disease. A Prospective Multicenter Follow-up Protocol With a Nested Randomized Controlled Trial of Physical Education Benefits - The SEDKID Study
Brief Title: SEDentary Lifestyle, Mortality and Major Adverse Clinical Outcomes in Chronic KIDney Disease
Acronym: SEDKID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: Satasairaala (Other); Vaasa Central Hospital, Vaasa, Finland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: T1451/2023
Record Dates: First submitted 2025-03-10; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: Chronic Kidney Disease; Cardiovascular Diseases; Frailty
Keywords: Chronic Kidney Disease; Cardiovascular Diseases; Renal Replacement Therapy; Frailty; Mortality; Hospitalisations; Exercise Program; Quality of Life; Emergency Department Visit; Major Adverse Cardiovascular and Cerebrovascular Events
MeSH Terms: conditions — Renal Insufficiency, Chronic; Cardiovascular Diseases; Frailty | interventions — Exercise; Dosage Forms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise Program (Experimental)
  Interventions: Behavioral: EXERCISE TRAINING WITH OR WITHOUT MEDICATION
- Standard of Care (No Intervention)

INTERVENTIONS:
Behavioral: EXERCISE TRAINING WITH OR WITHOUT MEDICATION — Single appointment with a registered physiotherapist educating the patient for rehabilitating physical training and exercise to be performed independently and regularly by the patient at home, minimum of three times a week, during the study period.
  Other Names: physical training education program
  Arms: Exercise Program

SUMMARY:
The goal of this study is to learn if a simple home exercise program can benefit patients with advanced chronic kidney disease. There is also an observational part of the study without an exercise program.

The study will record patients' mortality, cardiovascular events, emergency department visits, hospital stays, need for dialysis and 6 minutes walking distance. Also maximal oxygen uptake, quality of life and bone fractures are recorded and blood tests and X-rays analyzed. The prospective observational part of the study will investigate the link between cardiovascular and kidney health as well as exercise capacity and adverse outcomes.

DETAILED DESCRIPTION:
The prevalence of chronic kidney disease (CKD) and patients on maintenance dialysis is increasing, and affected patients are at elevated risk of premature death and adverse cardiovascular events.

Frailty is a term used to describe aging related attenuation of physical, mental, psychological and cognitive performance. Frailty is common in patients with CKD. Frailty is associated with increased mortality, hospitalization and falls in both the general population and in CKD.

Treatment of frailty is challenging due to its multidimensional nature and the old age and comorbidity of the affected patients. In spite these challenges, physical rehabilitation and training programs have been shown to successfully improve the prognosis of patients with CKD.

The investigators hypothesize that marked frailty is associated with a weak prognosis in spite renal replacement therapy and kidney transplantation. Because advanced predialysis stage CKD carries a high risk of adverse events and kidney transplants available are scarce, it is imperative to identify those elderly CKD stage 5 patients that benefit from initiating renal replacement therapy and those who are unlikely to benefit to avoid futile intensive treatment when it does not improve prognosis or quality of life. The investigators expect that the progression of frailty may up to a point be hindered using a simple physical exercise program that can be produced cost effectively to aid a large number of patients.

The trial aims to examine the benefits of an individual physical training education program in advanced CKD. In addition to the controlled trial setting the study examines the association between measures of frailty, physical and psychological capability assessed at study inclusion (baseline) and incident hospitalization, mortality, renal replacement therapy (RRT) and major adverse cardiovascular events during follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age >40 years
* Estimated glomerular filtration rate < 20ml/min/1.73m2 (CKD stage 4-5)
* Informed consent from the patient is received

Exclusion Criteria:

* Maintenance dialysis dependency before inclusion
* Pregnant women
* Patient's lack of commitment to follow-up
* Chronic or acute clinical condition with a prognosis less than 6 months
* Amputated lower limbs

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2025-02-21 (Actual); Primary Completion 2031-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Hospitalisations | 1 year, 2 years, 3 years, 5 years, 31 Dec 2031
Mortality | 1 year, 2 years, 3 years, 5 years, 31 Dec 2031
Major Adverse Cardiovascular or Cerebrovascular Event (MACCE) | 1 year, 2 years, 3 years, 5 years, 31 Dec 2031
Emergency Department Visits | 1 year, 2 years, 3 years, 5 years, 31 Dec 2031
6-minute Walking Test Distance | 1 year, 2 years, 3 years, 5 years, 31 Dec 2031
Renal Replacement Therapy | 1 year, 2 years, 3 years, 5 years, 31 Dec 2031
  start of dialysis or kidney transplantation
Compliance to the home training program | 1 year, 2 years, 3 years, 5 years, 31 Dec 2031
  Compliance of the intervention group assessed at every clinical control visit and tri-monthly by telephone.

SECONDARY OUTCOMES:
Maximal oxygen uptake in the exercise stress test | 1 year, 2 years, 3 years, 5 years, 31 Dec 2031
  Measured by spiroergometry (adjusted by body weight ml/kg/min)
Change in Quality of life | 1 year, 2 years, 3 years, 5 years, 31 Dec 2031
  Measured by RAND-36 questionnaire (8 domains and 2 composite scores, scale 0-100, higher score indicating better quality of life)
Bone fractures | 1 year, 2 years, 3 years, 5 years, 31 Dec 2031
  Number of participants with incident fractures, total number of fractures

CONTACTS AND LOCATIONS:
Overall Officials: Tapio Hellman, MD, PhD, Principal Investigator — Turku University Hospital and University of Turku; Mikko J Järvisalo, MD, PhD, Principal Investigator — Satasairaala Hospital, Wellbeing Services County of Satakunta
Locations (3):
- Finland (3):
  - Satasairaala Hospital, Pori
  - Turku University Hospital, Turku
  - Vaasa Central Hospital, Vaasa